CLINICAL TRIAL: NCT00526201
Title: Arthritis Benefits of a Physical Activity Program in West Virginia: Evaluation of EnhanceFitness
Brief Title: Help Arthritis With Exercise in West Virginia
Acronym: HARE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jennifer Hootman (U.S. Federal Agency)
Collaborators: West Virginia University (Other)
Responsible Party: Sponsor-Investigator, Jennifer Hootman, Epidemiologist, Centers for Disease Control and Prevention
Organization: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDC-NCCDPHP-AAMC-0944; AAMC-0944
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Arthritis
Keywords: Arthritis; Osteoarthritis; Rheumatoid Arthritis; Fibromyalgia; Lupus
MeSH Terms: conditions — Arthritis; Osteoarthritis; Arthritis, Rheumatoid; Fibromyalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Experimental): Subjects will be randomized to exercise (12 week EnhanceFitness class) or a wait-list control group.
  Interventions: Behavioral: 12-weeks EnhanceFitness
- Control (Other): Wait-list control group will receive intervention after 12-weeks.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: 12-weeks EnhanceFitness — EnhanceFitness class for 12 weeks, 3 times per week for 1 hour sessions.
  Arms: Exercise
Behavioral: Control — Participants randomized to the wait-list control group will continue their regular activities for 12 weeks and then be offered the exercise intervention (EnhanceFitness).
  Arms: Control

SUMMARY:
The purpose of this project is to determine if an evidence-based, community-delivered physical activity program, EnhanceFitness, yields benefits for participants with arthritis. The 3-year project will: 1) conduct a meta-analysis of community-based exercise programs for adults, 2) implement and evaluate the EnhanceFitness program in West Virginia using a randomized, controlled (wait list) design, and 3) disseminate the results to community and public health partners. It is anticipated that participation in the EnhanceFitness program will result in reduced pain, improved physical function and physical activity levels for adults with arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Any type of self-reported, doctor-diagnosed arthritis

Exclusion Criteria:

* Any co-existing conditions where exercise is a contraindicated
* Impaired cognitive status
* Non-ambulatory

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2009-05; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Pain Severity | 8 months
Physical activity level | 8 months
Physical Function | 8 months

SECONDARY OUTCOMES:
Health-related quality of life | 8 months
Arthritis self-efficacy | 8 months
Self-efficacy for exercise | 8 months
Exercise perceptions | 8 months
Social support | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Dina L Jones, PT, PHD, Principal Investigator — West Virginia University; Jennifer M Hootman, PhD, Study Director — Centers for Disease Control and Prevention
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States

REFERENCES:
- [Derived] Jones DL, Eicher JL, Fang W, Hootman JM. Effectiveness and Implementation of an EnhanceFitness Physical Activity Intervention Specifically in Adults With Arthritis: A RE-AIM Evaluation. Gerontologist. 2024 Jul 1;64(7):gnad157. doi: 10.1093/geront/gnad157. PMID 38051008